CLINICAL TRIAL: NCT00923000
Title: Herb Drug Interaction of Traditional Chinese Herb and Commonly Used Drugs
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Shung-Tai Ho/Professor, Tri-Service General Hospital
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DDI-001; TSGHIRB096-02-015-A
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2009-06-19 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: Herb Drug; volunteers
MeSH Terms: interventions — Nalbuphine; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Nubian with Long dan xie gan tang 3g (Experimental)
  Interventions: Drug: Nubian with Long dan xie gan tang
- Nalbuphine (Active Comparator)
  Interventions: Drug: Nalbuphine
- Morphine (Active Comparator)
  Interventions: Drug: Morphine
- Morphine with Long dan xie gan tang (Experimental)
  Interventions: Drug: Morphine with Long dan xie gan tang
- Nubian with Long dan xie gan tang 3g tid (Experimental)
  Interventions: Drug: Nalbuphine with Long dan xie gan tang

INTERVENTIONS:
Drug: Nalbuphine — Nalbuphine 10mg with oral administration
  Arms: Nalbuphine
Drug: Morphine — Morphine 10mg with oral administration
  Arms: Morphine
Drug: Morphine with Long dan xie gan tang — Morphine 10mg with oral administration
  Arms: Morphine with Long dan xie gan tang
Drug: Nalbuphine with Long dan xie gan tang — Nalbuphine 10mg with Long dan xie gan tang 3g tid with oral administration
  Arms: Nubian with Long dan xie gan tang 3g tid
Drug: Nubian with Long dan xie gan tang — Nalbuphine 10mg with Long dan xie gan tang 3g with oral administration
  Arms: Nubian with Long dan xie gan tang 3g

SUMMARY:
The purpose of this study was to investigate a possible response to nalbuphine (Nubian) and morphine with traditional Chinese herbs in healthy volunteers.

DETAILED DESCRIPTION:
This study is a single center and open-label design to investigate the pharmacokinetic properties of Nubian, Nubian traditional Chinese herb combination dosage after single oral with oral administration, or morphine, morphine traditional Chinese herb combination dosage after single oral administration in healthy volunteers under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy adult subjects between 20-40 years of age
* Body weight within 80-120% of ideal body weight
* Acceptable medical history, physical examination and clinical laboratory determinations

Exclusion Criteria:

* Recent history of drug or alcohol addiction or abuse
* Donating greater than 150 ml of blood within two months prior to Period I
* Taking any prescription medication or any nonprescription medication within 14 days prior to Period I doing
* Receiving any investigational drug within 30 days prior to Period I dosing
* Taking any drug known to induce or inhibit hepatic drug metabolism within 30 days prior to the beginning of the study
* Any clinically significant diseases
* History of allergic response to nalbuphine or related drugs and traditional Chinese herbs

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The pharmacokinetic parameters | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Tai Ho, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan